CLINICAL TRIAL: NCT01372943
Title: A Study Using "Synthetic Stool" or Pure Cultures of Probiotic Intestinal Bacteria From Healthy Donor Stool That Can be Used as an Enema to Replace the Use of Stool Transplant, for Treatment of Recurrent and Refractory CDI
Brief Title: Harnessing the Healthy Gut Microbiota to Cure Patients With Recurrent C. Difficile Infection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Research priorities and focus have shifted
Sponsor: Queen's University (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Dr. Mark Ropeleski, Physician, Queen's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMED 1318-10
Record Dates: First submitted 2011-06-08; First posted 2011-06-14 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Clostridium Difficile Infection
Keywords: Clostridium difficile; recurrent; infection
MeSH Terms: conditions — Clostridium Infections; Recurrence; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- synthetic stool (Experimental): "synthetic stool" or pure cultures of probiotic intestinal bacteria from healthy donor stool that can be used as an enema to replace the use of stool transplant, for treatment of recurrent and refractory CDI
  Interventions: Biological: "synthetic stool" or pure cultures of probiotic intestinal bacteria

INTERVENTIONS:
Biological: "synthetic stool" or pure cultures of probiotic intestinal bacteria — "synthetic stool" or pure cultures of probiotic intestinal bacteria from healthy donor stool that can be used as an enema to replace the use of stool transplant, for treatment of recurrent and refractory CDI

SUMMARY:
CDI (Clostridium difficile infection) causes diarrheal illness and can cause colitis which may be fatal. A patient being treated for CDI has a 10-25% chance of developing relapse. Recurrent CDI is on the rise. There are few options available to treat recurrent CDI. "Stool transplant" (infusing donor stool into the intestine of the recipient), is not very palatable to either patient or medical personnel. The investigators will isolate intestinal bacteria from donor stool and use this purified mixture of donor bacteria instead of stool transplant. The investigators hypothesize that this cleaner mixture of purely isolated intestinal bacteria from a healthy donor would be equally effective as conventional fecal bacteriotherapy, which uses donor stool. The use of this prepared mixture of aerobic and anaerobic organisms, or probiotic approach, is based on the same principle of fecal flora reconstitution. However our approach would provide a more controlled, reproducible, cleaner and more aesthetically acceptable method of administration, and from a patient safety perspective, would also be a safer strategy than using freshly defecated donor fecal matter.

ELIGIBILITY:
Inclusion Criteria:

* patients with recurrent CDI that have failed standard therapy

Exclusion Criteria:

* critically ill patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-01; Primary Completion 2017-01 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
number of participants cured of CDI | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Petrof, MD, Principal Investigator — Kingston Health Sciences Centre
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada

REFERENCES:
- [Derived] Petrof EO, Gloor GB, Vanner SJ, Weese SJ, Carter D, Daigneault MC, Brown EM, Schroeter K, Allen-Vercoe E. Stool substitute transplant therapy for the eradication of Clostridium difficile infection: 'RePOOPulating' the gut. Microbiome. 2013 Jan 9;1(1):3. doi: 10.1186/2049-2618-1-3. PMID 24467987